CLINICAL TRIAL: NCT06019078
Title: Continuous Processed Neurological Monitor to Guide the Management of Sedation for Patients Receiving Mechanical Ventilation: a Prospective Observational Study to Test the Effects on Delirium, Days on a Ventilator, and Post-Intensive Care Syndrome.
Brief Title: pEEG Monitoring Effect on Delirium, Ventilator Days, and PICS
Status: Completed | Type: Observational
Sponsor: Fraser Health (Other)
Collaborators: University of Victoria (Other)
Responsible Party: Sponsor
Other Study IDs: H23-01671
Record Dates: First submitted 2023-08-14; First posted 2023-08-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness; Post Intensive Care Unit Syndrome; Post Intensive Care Syndrome; Mechanical Ventilation Complication; Delirium; Sedative-Related Disorders; Subsequent Encounter; Analgesia
Keywords: criticial illness; post intensive care unit syndrome; post intensive care syndrome; mechanical ventilation complication; delirium
MeSH Terms: conditions — Critical Illness; postintensive care syndrome; Delirium; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: Patients admitted to participating ICUs who meet inclusion criteria monitored by 4 channel pEEG.
  Interventions: Device: SedLine
- Retrospective Cohort: Patients admitted to participating ICUs who meet inclusion criteria not monitored by 4 channel pEEG.

INTERVENTIONS:
Device: SedLine — Continuous 4 channel processed neurological monitor
  Groups: Prospective Cohort

SUMMARY:
The goal of this multi-site observational study is to compare delirium rates, days on mechanical ventilation, and Post Intensive Care Syndrome (PICS) rates in adult Intensive Care Unit (ICU) patients. The study will examine patients whose sedation and analgesia infusion titration is managed with both Richmond Agitation and Sedation Scale (RASS) and Processed Electroencephalography (pEEG) monitoring vs patients who receive RASS monitoring alone.

The main questions are:

* Compared to RASS monitoring method alone, does the use of 4 channel pEEG monitor in conjunction with RASS to guide the management of sedation and analgesic in patients who are ventilated reduce the average number of delirium days, measured by Intensive Care Delirium Screening Checklist (ICDSC)?
* To determine when compared to RASS monitoring alone if the use of 4 channel pEEG monitor in conjunction with RASS to guide the management of Intravenous (IV) sedation and analgesia in ventilated patients reduces the days a patient spends on a mechanical ventilator when compared to RASS only monitoring from retrospective data.
* To determine when compared to RASS monitoring method alone, does the use of 4 channel pEEG monitor in conjunction with RASS experience lower doses of sedation and analgesia infusions?
* To determine when compared to RASS monitoring method alone, does the use of 4 channel pEEG monitor in conjunction with RASS experience less incidence and duration of PICS?

DETAILED DESCRIPTION:
The purpose of this study is to determine the impact of using a 4 channel pEEG monitor to guide sedation and analgesia management in conjunction with RASS in ventilated patients in the ICU on length of time patients experience delirium, number of days patients spend on a ventilator, and incidence of PICS in these same patients.

Participants who are on a mechanical ventilator and on IV sedation or analgesia will be placed on a pEEG monitor on admission to ICU.

Participants will complete a battery of test at discharge, one month post discharge, and three months post discharge to assess for PICS.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to ICU
2. Receive mechanical ventilator support during ICU stay
3. Require IV sedation or analgesic while ventilated
4. Discharged home from the hospital
5. Use of pEEG for sedation or analgesic titration
6. Able to read and speak English
7. Mechanically ventilated greater than 48 hours
8. Aged 17 years +1 day or greater
9. Consent to participate
10. Participants need a computer with a keyboard, internet access, and email access for the questionnaires and assessment and be able to use computer and internet.

Exclusion Criteria:

1. Deceased during hospitalization
2. Intubated at a hospital not included within the study > 12 hours
3. Discharge to rehabilitation facility, long term care, or other outpatient setting
4. Inability to provide informed consent
5. Currently enrolled in any other research study involving drugs or devices
6. Is unable to be screened for delirium during ICU admission.

Ages: 17 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult medical and surgical ICU patients .
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Delirium | For the time the patient remains in ICU until discharge from ICU. Average length of stay in ICU is 7 days.
  Measured by Intensive Care Delirium Screening Checklist (ICDSC). The items include the assessment of: (1) consciousness ( deep sedation/coma, agitation, normal wakefulness, or light sedation); (2) inattention; (3) disorientation; (4) hallucination, delusion, or psychosis; (5) psychomotor agitation or retardation; (6) inappropriate speech or mood; (7) sleep-wake cycle disturbances; and (8) fluctuation of symptomatology. The maximum score is eight; scores of ≥4 indicate the presence of delirium and score zero is indicate not in delirium. Each item is scored 0-8.

SECONDARY OUTCOMES:
Days of Mechanical Ventilation | From the date of intubation until extubation in ICU. Average length of mechanical ventilation is 7 days.
  Measured at ICU discharge, measured as half days.
Sedation Infusions (Propofol and/or Midazolam) | Measured every 4 hours while the patient remains on the infusion in ICU. Average length of time spent on a sedation infusion is 5 days.
  Rates and dosages of sedation infusions
Combined Sedation and Analgesia Infusions (Dexmedetomidine and/or Ketamine) | Measured every 4 hours while the patient remains on the infusion in ICU. Average length of time spent on a combined sedation and analgesic infusion is 3 days.
  Rates and dosages of sedation and analgesic infusions
Analgesia Infusions (Fentanyl, Morphine, and/or Hydromorphone) | Measured every 4 hours while the patient remains on the infusion in ICU. Average length of time spent on an analgesic infusion is 5 days.
  Rates and dosages of analgesic infusions
Computerized Neurocognitive Screening Vital Signs | At hospital discharge (4 days +/- 1) average length of stay in hospital 5-90 days, 1 month post discharge, 3 months post discharge
  CNS Vital Signs (CNSVS) is a computerized neurocognitive test battery that was developed as a routine clinical screening instrument. It is comprised of seven tests: verbal and visual memory, finger tapping, symbol digit coding, the Stroop Test, a test of shifting attention and the continuous performance test. Standard Scores are normalized from raw scores and present an age matched score relative to other people in a normative sample. CNS Vital Signs standardized have a mean of 100 and a standard deviation is 15. Higher scores are always better.
Hospital Anxiety and Depression Scale | At hospital discharge (4 days +/- 1) average length of stay in hospital 5-90 days, 1 month post discharge (6 days +/- 1) , 3 months post discharge (6 days +/- 1)
  The questionnaire comprises seven questions for anxiety and seven questions for depression. For both scales, scores of less than 7 indicate non-cases, score of 8-10 mild case, 11-14 moderate case, and 15-21 severe case.
Impact of Events Scale-Revised | At hospital discharge (4 days +/- 1) average length of stay in hospital 5-90 days, 1 month post discharge (6 days +/- 1) , 3 months post discharge (6 days +/- 1)
  The IES-R is a validated 22-item self-report scale measuring psychological stress reactions after a major life or traumatic event.1-3Items are rated with reference to the past 7 days on a 5-point scale, ranging from 0 to 4. Three subscale scores are calculated by taking the mean of the item responses: Intrustion (8 items), Avoidance (8 items), and Hyperarousal (6 items). The total score is similarly computed by taking the mean of all 22 items. All scores range from 0 to 4, with higher scores indicating higher event-related distress. Internal consistency estimates(Cronbach's alpha) for all scores range between 0.79 to 0.92.
EuroQol-5D-5L | At hospital discharge (4 days +/- 1) average length of stay in hospital 5-90 days, 1 month post discharge (6 days +/- 1) , 3 months post discharge (6 days +/- 1)
  Health related quality of life questionnaire EuroQol-5D-5L is used. Five levels are score in 5 dimensions. It is scaled from 0 to 100%. A higher score indicates a higher quality of life.
Suppression Ratio | From the time pEEG monitoring is initiated until it is discontinued. Average length of time spent on a pEEG monitor is 5 days.
  Percentage of time the patient's brain is in burst suppression. Scored on a numerical scale 0-100%. A lower percentage is better.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona E Howarth, Principal Investigator — Fraser Health
Locations (1):
- Abbotsford Regional Hospital, Abbotsford, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.